CLINICAL TRIAL: NCT06783985
Title: Clinical Application of Carbon Nanoparticles in Lymph Node Tracing and Surgery Guiding of Colorectal Cancer
Acronym: CNP-CRC
Status: Completed | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Bingjun Bai, Professor, Sir Run Run Shaw Hospital
Other Study IDs: SirRRSH-CNP-CRC
Record Dates: First submitted 2025-01-08; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer
Keywords: carbon nanoparticle; colorectal cancer; lymph node
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CNP group: Every patient received endoscopic injection of 0.5 ml CNP suspension (Chongqing LUMMY Pharmaceutical Co., Chongqing, China) into submucosal layer at one point, at the lower margin of the tumor. All patients subsequently underwent laparoscopic or robotic radical resection with D3 LN dissection. Tumor tissue and LNs s were isolated from surgical specimen by the same pathologist. LNs dissection and harvest were on the basis of the Japanese classification of colorectal carcinoma.

SUMMARY:
This trial aims to clarify the relationship between carbon nanoparticles labeled lymph nodes and lymph node metastasis in different lymph node regions of colorectal cancer, and to clarify the application value of carbon nanoparticles in lymph node dissection in colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of colorectal cancer;
2. endoscopic injection of CNP suspension preoperatively
3. planned radical resection of colorectal cancer
4. older than 18 years of age

Exclusion Criteria:

(a) emergency surgery;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted in Sir Run Run Shaw Hospital, Zhejiang University School of Medicine. Patient information and samples were obtained from patients undergoing radical resection of colorectal cancer in the colorectal surgery department of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
The relationship between carbon nanoparticle stained lymph nodes and metastatic lymph nodes | From enrollment to the pathology report at 2 weeks

SECONDARY OUTCOMES:
Carbon nanoparticle stained lymph nodes from different lymph node groups. | From enrollment to the pathology report at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol